CLINICAL TRIAL: NCT04388124
Title: VASCULAR AND RENAL IMPACT OF ENDOTHELIN-1 RECEPTOR BLOCKADE IN PATIENTS WITH RESISTANT ARTERIAL HYPERTENSION
Acronym: ENDOTHELIN-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/350/HP
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Resistant Hypertension
Keywords: endothelin-1
MeSH Terms: interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Modification of the pharmaceutical form, removal from the primary packaging and repackaging-> tablet of Bosentan will be encapsuled. The pharmaceutical form of placebo and bosentant will be identical
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patient will receive placebo for 56 days: 2 capsules of 62.5 mg per day for 27 days +/-1 day, 2 capsules of 125 mg per day for 27 days +/-1 day.
  Interventions: Drug: Placebo
- Bosentan (Experimental): Patient will receive Bosentan for 56 days: 2 capsules of 62.5 mg per day for 27 days +/-1 day, 2 capsules of 125 mg per day for 27 days +/-1 day.
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — vascular assesment Clinical exam urinary analysis blood results natriuresis and measured glomerular filtration rate
  Arms: Bosentan
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The management of patients with resistant arterial hypertension, who are characterized by a very high cardiovascular risk, remains a major therapeutic issue. The use of endothelin-1 (ET-1) receptor antagonists, in addition to lowering blood pressure, may also improve endothelial function in these patients. The objective of this study is to assess the vascular impact of an ET-1 receptor antagonist on vascular function and systemic and central hemodynamics in patients with resistant arterial hypertension and ensure their good renal tolerance.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 80 years old
* Patients with resistant hypertension defined according to the criteria recognized by the French Society of Hypertension (SFHTA): arterial pressure greater than or equal to 140 and / 90 mm Hg under triple antihypertensive therapy at optimal dose comprising at least one diuretic pendant at less than 4 weeks.
* Patients with resistant hypertension confirmed by self-measurement (≥135 / 85 mmHg on average) or by ambulatory blood pressure measurement (mean of 24h ≥130 / 80 mmHg).
* Hemoglobin level ≥ 12 g / dL
* For women of childbearing potential, reliable methods of contraception (as defined by the WHO-Pearl Index) should be used (hormonal contraception should not be the only contraceptive method used during bosentan treatment).
* For postmenopausal women: confirmatory diagnosis (non-medically induced amenorrhea for at least 12 months and age greater than 45, before the inclusion visit)
* Patient who read and understood the newsletter and signed the consent form
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patients with hypertension
* Patients with secondary arterial hypertension other than sleep apnea syndrome or chronic renal failure stage 2 or 3.
* Patients with hypertension greater than or equal to 180 and / or 110mmHg
* Chronic renal failure stage 4 and 5 (defined by DFG CKD-EPI <30 ml / min / 1,73m²)
* Renal transplant patient XML File Identifier: CEyMau8sPo+QFyOLD1ZEY3ZGFow= Page 11/22
* Orthostatic hypotension (decreased SBP> 20mmHg and / or DBP> 10mmHg occurring within 3 minutes of standing).
* Contra-indication to NATISPRAY 0.30 mg / dose, oral spray solution (including nitrate hypersensitivity) in accordance with the NATISPRAY

SPC:

* shock, severe hypotension,
* in combination with sildenafil
* obstructive cardiomyopathy,
* inferior court inferior myocardial infarction with right ventricular extension, except in case of evidence of left ventricular failure,
* intracranial hypertension,

  • Contra-indication to BOSENTAN MYLAN 62.5 mg and 125 mg filmcoated tablets:
* Hypersensitivity to the active substance or to any of the excipients listed in the SPC Moderate to severe hepatic insufficiency corresponding to class B or C of the Child-Pugh classification
* Serum levels of liver aminotransferases, ASAT and / or ALAT> 3 times the upper limit of normal at start of treatment (results less than 3 months old).
* Association with ciclosporin A

  * Known allergy to cellulose
  * Patients treated with: tacrolimus or sirolimus, fluconazole or other CYP2C9 or CYP3A4 inhibitors, glibenclamide, rifampicin, antiretroviral drugs including lopinavir + ritonavir, warfarin, simvastatin, ketoconazole, epoprostenol, sildenafil and digoxin
  * Pregnant, breastfeeding woman, or woman of childbearing potential not using reliable methods of contraception (hormonal contraception should not be the only contraceptive method used during bosentan treatment) or no proven reliable effective contraception;
  * Person deprived of liberty by an administrative or judicial decision or person placed under the protection of justice, under tutorship or curatorship
  * Patient participating or having participated in the 4 weeks prior to inclusion in a clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
assess the effect of ET-1 receptor antagonist administration during 8 weeks on endothelial function in patients with resistant hypertension. | through study completion, an average of 22 months
  8-week change in amplitude of endothelium-dependent radial artery dilatation with sustained increase in blood flow

SECONDARY OUTCOMES:
assess the effect of the administration of an ET-1 receptor antagonist during 8 weeks on systemic and central hemodynamics | through study completion, an average of 22 months
  8 week change in peripheral and central arterial pressures and arterial stiffness
assess the effect of the administration of an ET-1 receptor antagonist during 8 weeks on local concentrations of endothelial factors during a sustained increase of the blood flow | through study completion, an average of 22 months
  8-week change in local concentrations of NO, EETs and ET-1 with sustained increase in blood flow
assess the effect of the administration of an ET-1 receptor antagonist during 8 weeks on the renal function of patients with resistant hypertension. | through study completion, an average of 22 months
  Variation in 8 weeks of natriuresis and measured glomerular filtration rate (DTPA labeled by the technetium 99m)